CLINICAL TRIAL: NCT06810167
Title: An Open-label, Single Center Study Assessing Tenapanor as a Non-CFTR-mediated Treatment of CF-related Constipation in People With CF.
Brief Title: Assessing Tenapanor as a Treatment of CF-related Constipation.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ardelyx (Industry)
Responsible Party: Principal Investigator, Christopher Velez, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002058
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis; Constipation
Keywords: Constipation; Cystic Fibrosis; CFrC
MeSH Terms: conditions — Cystic Fibrosis; Constipation | interventions — tenapanor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cystic fibrosis patients with CF-related constipation (Experimental)
  Interventions: Drug: Tenapanor

INTERVENTIONS:
Drug: Tenapanor — CF patients with CFrC will ingest one 50 mg tablet of tenapanor twice daily for 4 weeks.

SUMMARY:
Tenapanor is the newest FDA-approved drug for IBS with constipation (IBS-C). This study seeks to understand tenapanor as a treatment for cystic fibrosis-related constipation (CFrC) in CF patients. Participants will ingest one 50 mg tablet of tenapanor, twice daily, for a 4-week treatment period. They will also complete three questionnaires, the PAC-SYM, PAC-QoL, and IBS-SSS, and daily diaries to characterize GI symptom burden and spontaneous bowel movement (SBM) frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Having confirmed cystic fibrosis (either by sweat chloride or genetic testing)
2. Meeting criteria for CFrC

   Must include 2 of the following, with or without abdominal pain for at least 3 months, with symptom onset at least 6-months prior:
   * Straining in at least 25% of defecations
   * Bristol Stool Scale 1-2 more than 25% of defecations (change in stool form)
   * Sensation of incomplete evacuation more than 25% of defecations
   * Sensation of anorectal obstruction/blockage more than 25% of defecations
   * Manual disimpaction/manipulation of pelvic floor to facilitate more than 25% of defecations
   * Fewer than 3 spontaneous bowel movements weekly (change in stool frequency)
   * Loose stools rarely present without the use of laxatives
3. Willingness to avoid major dietary or lifestyle changes during study.

Exclusion Criteria:

1. Use of any antibiotic to treat infection within the 4-weeks prior to study initiation (stable azithromycin dosed 3-times weekly for lung function is to be allowed)
2. Inability to discontinue standing bowel regimen (including fiber, stool softener, as well as either osmotic or stimulant laxative, pro-kinetic serotonergic agents, or other therapy) 2-weeks prior to study drug initiation (with ability to use osmotic laxative therapy as rescue therapy only).
3. Severe CFrC as determined by study team
4. Prior tenapanor usage
5. Hospitalization within 4-weeks prior to study initiation.
6. DIOS within 4-weeks prior to study initiation.
7. Other known/suspected mechanical obstruction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase in SBM frequency | Patients will record SBM frequency over the 4-week treatment period.
  There will be a statistically significant increase in spontaneous bowel movement frequency (SBM) in cystic fibrosis patients with CF-related constipation receiving tenapanor.

SECONDARY OUTCOMES:
Change in PAC-SYM questionnaire score | Patients will complete the PAC-SYM at -2 weeks, 0 weeks, 2 weeks, and 4 weeks.
  There will be a change (with use of descriptive statistics) in bowel symptoms characterized by the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire with tenapanor administration. PAC-SYM is a PRO previously used to examine constipation in pwCF. A decreased score corresponds to improvement of bowel symptoms.
Change in PAC-QOL questionnaire score | Patients will complete the PAC-QOL at -2 weeks, 0 weeks, 2 weeks, and 4 weeks.
  There will be a change (with use of descriptive statistics) in bowel symptoms characterized by the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire with tenapanor administration. PAC-QOL is a PRO previously used to examine constipation in pwCF. A decreased score corresponds to improvement of bowel symptoms.
Change in IBS-SSS questionnaire score | Patients will complete the IBS-SSS at -2 weeks, 0 weeks, 2 weeks, and 4 weeks.
  There will be a 50-point change in the Irritable Bowel Syndrome Scoring System - IBS-SSS (in line with recent bowel distress related literature Ford AC, Wright-Hughes A, Alderson SLet al Lancet 2023) in pwCF and CFrC receiving tenapanor.

CONTACTS AND LOCATIONS:
Overall Officials: Christoher D Velez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No